CLINICAL TRIAL: NCT03099525
Title: Treatment Outcome and Prognostic Factors for RA Patients With Interstitial Lung Disease
Brief Title: Treatment Outcome and Prognostic Factors for Rheumatoid Arthritis (RA) Patients With Interstitial Lung Disease (ILD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yoon-Kyoung Sung, Associate professor, Hanyang University
Other Study IDs: HUHRD-SPE-16-08
Record Dates: First submitted 2017-01-26; First posted 2017-04-04 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA-ILD: Patients who are diagnosed with ILD. No intervention in this study.
  Interventions: Other: ILD
- RA-non ILD: Patients who are not diagnosed with ILD. No intervention in this study.
  Interventions: Other: ILD

INTERVENTIONS:
Other: ILD — This is an observational study without any intervention.

SUMMARY:
The objectives of this single center, prospective, non-interventional cohort is to understand patient characteristics, general treatment patterns, effectiveness/safety of conventional disease modifying antirheumatic drug (DMARD) and biologic DMARD treatments in rheumatoid arthritis patients with ILD in the real-world setting

DETAILED DESCRIPTION:
Primary objective

: Comparison of prognosis between RA-ILD and RA-non ILD patients

Secondary objectives

1. Identification of the prognostic factors or aggravation factors of ILD in RA-ILD patients
2. Identification of the association between ILD and autoantibody profiles in RA-ILD patients
3. Comparison of RA disease activity control between RA-ILD and RA-non ILD patients using disease activity score (DAS)28-erythrocyte sedimentation ratio (ESR), DAS28 C-reactive protein (CRP), simple disease activity index (SDAI) and clinical disease activity index (CDAI)
4. Comparison of biologic and non-biologic DMARD treatment response in RA-ILD patients using disease activity parameters

The study population will be adult RA patients who have checked a chest computed tomography (CT) scan within 2 years of enrollment. No additional visits or laboratory tests will be done outside the routine clinical practice for RA-non ILD patients. For RA-ILD patients, high resolution computed tomography (HRCT), pulmonary function test (PFT) and 6-min walk test will be examined annually to identify the progression of ILD. Selection of medication including conventional DMARDs, biologic DMARDs, glucocorticoid, and inhaler, dosing and treatment duration are at the discretion of the investigator.

ELIGIBILITY:
A. Inclusion Criteria:

* Patients who satisfy the 1987 American college of rheumatology (ACR) or 2010 ACR/EULAR classification criteria for RA adult patients
* Patients who are more than 19 years old
* Patients who have checked chest CT scanning within 2 years
* Patients who provide a written consent of participating in this study

B. Exclusion Criteria:

* Patients who are aged under 19 years old
* Patients who are pregnant
* Patients who dose not provide a written consent of participating in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients diagnosed with RA with normal chest CT result within 2 years of clinical visit.
  Korean patients diagnosed with RA-ILD with chest CT results indicating ILD within 2 years of clinical visit.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  Comparison of prognosis such as mortality between RA-ILD and RA-non ILD

SECONDARY OUTCOMES:
Pulmonary function test | 5 years
  Identify aggravation factors for RA-ILD
DAS28(Disease Activity Score in 28 joint) | 5 years
  Comparison of RA disease activity control between RA-ILD and RA-non ILD using Disease Activity Score(DAS28)
SDAI(Simple Disease Activity Index) | 5 years
  Comparison of RA disease activity control between RA-ILD and RA-non ILD using Simple Disease Activity Index(SDAI)
CDAI(Clinic Disease Activity Index) | 5 years
  Comparison of RA disease activity control between RA-ILD and RA-non ILD using Clinic Disease Activity Index(CDAI)
Change of DAS28 | 5 years
  Comparison of biologic and non-biologic DMARDs treatment response in RA patients

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Kyoung Sung, MD,PhD,MPH, Principal Investigator — Hanyang University Hospital for Rheumatic Diseases
Locations (1):
- Hanyang University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Cho SK, Song YJ, Kang J, Jeong SA, Kim HW, Choi CB, Kim TH, Jun JB, Bae SC, Yoo DH, Lee H, Park DW, Sohn JW, Yoon HJ, Hong SJ, Yoo SJ, Choi YW, Lee Y, Kim SH, Sung YK. Clinical characteristics of rheumatoid arthritis patients with interstitial lung disease: baseline data of a single-center prospective cohort. Arthritis Res Ther. 2023 Mar 17;25(1):43. doi: 10.1186/s13075-023-03024-8. PMID 36932433